CLINICAL TRIAL: NCT05205278
Title: Effect of Progressive Isolated Core Stability Training on Upper Extremity Physical Performance in Adolascent Female Volleyball Athletes
Brief Title: Effect of Progressive Isolated Core Stability Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUT 12/57
Record Dates: First submitted 2021-12-05; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-12

CONDITIONS: CORE STABILITY; Upper Extremity; Physical Performance
Keywords: athlete; exercise; muscle strength; flexibility
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Forty-two adolescent female volleyball athletes (16.0±1.4 years) were randomly divided into two groups. Group 1 was the training group and, in addition to the routine volleyball training programmes, underwent an 8-week (3 days/week) progressive core stability training programme. Group 2 was the control group and only did routine volleyball training, with no core stability training.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training group (Experimental): Group 1 (n=21) was the training group and, in addition to the routine volleyball training programmes, an 8-week (3 days/week) progressive core stability training programme was applied.
  Interventions: Other: exercise training
- control group (No Intervention): Group 2 (n=21) was the control group, and they only engaged in routine volleyball training: no core stability training was given.

INTERVENTIONS:
Other: exercise training — The core stability training programme was performed 3 days per week over an 8-week period, and each training session lasted approximately 50 minutes.We created a special programme for our study based on the literature; the core stability training programme was divided into 3 phases: easy(1-2 weeks), moderate(3-5 weeks) and difficult(6-8 weeks In the easy phase(phase1), the athlete was intended to gain sensorimotor control that would ensure the smoothness of the neutral spine during slow movements. The participants learned the hallowing technique and how to use this technique while doing core exercises. In the moderate phase(phase2), muscular neural adaptation and neuromuscular facilitation were targeted with the transition to high threshold strength training.In the last, difficult, phase(phase3), subconscious control of movement was taught using combined movement patterns with the aim of transitioning to functional positions and activities.
  Arms: training group

SUMMARY:
Forty-two adolescent female volleyball athletes (16.0±1.4 years) were randomly divided into two groups. Group 1 was the training group and, in addition to the routine volleyball training programmes, underwent an 8-week (3 days/week) progressive core stability training programme. Group 2 was the control group and only did routine volleyball training, with no core stability training.

Main outcome measures: Shoulder IR and ER strength, medicine ball throw (MBT), modified push up (MPU) and closed kinetic chain (CKC) upper extremity stability tests were used to evaluate physical performance.

DETAILED DESCRIPTION:
Most studies have focused on the effects of core stability training on injury prevention and physical performance for the lower extremities . However, little is known about its effect on upper extremity performance. Previous studies suggest that core strengthening could enhance upper extremity physical performance because it might lead to more efficient use of the extremity muscles . Core weakness in overhead athletes with shoulder pain. Insufficient power generation by the core muscles might overload the shoulder girdle to compensate for altered biomechanics during throwing, and this overload made the shoulder prone to sport injuries. A systematic review has suggested, however, that isolated core stability training cannot be the primary component of athletic performance enhancement and that the variability in exercise training protocols, testing methods, study population and sample size among the available studies leads to difficulties in understanding whether or not core stability training enhances physical performance.

There has been no study in the literature investigating the effect of progressive isolated core stability training on upper extremity performance in adolescent overhead athletes. This study therefore sought to investigate the effects of progressive isolated core stability training on shoulder internal (IR) and external rotator (ER) strength and upper extremity physical performance in female adolescent volleyball players. Hypothesized that core stability training would enhance shoulder rotator strength and upper extremity physical performance in these athletes.

ELIGIBILITY:
Inclusion Criteria:

- be between the ages of 12 and 16, enrolled in a similar training program and agree to participate in the study

Exclusion Criteria:

* Having any surgery / serious pathology of the spinal column,
* Have had a lower / upper extremity injury in the last 3 months,
* Sports age is less than 5 years,
* Severe orthopedic / systemic discomfort during training,
* Absence from training for more than 3 sessions
* Family disapproval or reluctance to study
* Minimal Q-DASH score (0-25)

Ages: 12 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2013-03-15 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Shoulder Rotator Muscle Strength at 8 weeks. | before and after treatment (24 sessions, beginning and 8th. weeks)
  Isometric shoulder IR and ER strength was measured using a handheld dynamometer (Commander Power Track II, J-Tech, USA). The tests were performed with the athletes in a supine position. The shoulder was positioned at 45° abduction, the elbow was at 90° flexion and the forearm was in the neutral position. The supine position was chosen for the test to minimize compensatory movement of the body. At least one practice trial was given to the subjects to familiarize them with the feel of pushing against the dynamometer. Subjects were oriented to each desired action by the tester. The subject then performed the action until performed correctly.
Change from Baseline Upper Extremity Functional Tests at 8 weeks. | before and after treatment (24 sessions, beginning and 8th. weeks)
  The participants were positioned prone with hands shoulder width apart with the trunk held in a rigid straight position on the mat. Push-ups were performed through the full range of motion, as quickly as possible. Participants started the test with their elbows fully extended. They then flexed their elbows until the upper arm was parallel to the testing surface. The participants were instructed to limit head and trunk motion and to keep the trunk position straight. The number of push-ups completed in 30 seconds was recorded. Verbal encouragement was consistently given to all participants .
Change from CKC upper extremity stability test at 8 weeks. | before and after treatment (24 sessions, beginning and 8th. weeks)
  This test was performed in a modified push-up test position. There were two lines on the floor, 30 cm apart. The participants were instructed to move their hands back and forth from each line as many as possible for 15 seconds. The number of touches for each line was counted. The test was repeated 3 times, with a 2-minute rest between each trial and the average of the touches was calculated. The final score was calculated as the average number of touches/height
Change from MBT test at 8 weeks. | before and after treatment (24 sessions, beginning and 8th. weeks)
  The examiner used a marked line on the floor as the starting reference for this test. A mat was placed on the floor and the front of the mat was aligned with the reference line. The participants were instructed to tall kneel (90° knee flexion and neutral trunk position) on the front of the mat with the medicine ball (1.9 kg) held at their chest level against the chest wall. From this position the participants were instructed to throw the medicine ball, using a 2-handed chest pass technique, as far as they could. To minimize momentum, the participants were not allowed to rock back before beginning the throw. The first contact site of the ball was marked, and the throw distance was measured using tape. The test was repeated 3 times, and the average of the throw distances was calculated

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Tugba Kilic, Study Director — Ankara Yildirim Beyazıt University; Gülsah Basandac, Principal Investigator — Yeditepe University Department Of Physiotherapy And Rehabilitation; Gülcan Harput, Study Chair — Hacettepe University, Faculty of Physiotherapy and Rehabilitation; Volga Bayrakci Tunay, Study Chair — Hacettepe University, Faculty of Physiotherapy and Rehabilitation
Locations (1):
- Ankara Yildirim Beyazit University,Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bahr R, Reeser JC; Federation Internationale de Volleyball. Injuries among world-class professional beach volleyball players. The Federation Internationale de Volleyball beach volleyball injury study. Am J Sports Med. 2003 Jan-Feb;31(1):119-25. doi: 10.1177/03635465030310010401. PMID 12531768
- [Background] Reeser JC, Joy EA, Porucznik CA, Berg RL, Colliver EB, Willick SE. Risk factors for volleyball-related shoulder pain and dysfunction. PM R. 2010 Jan;2(1):27-36. doi: 10.1016/j.pmrj.2009.11.010. PMID 20129510
- [Background] Kibler WB, Press J, Sciascia A. The role of core stability in athletic function. Sports Med. 2006;36(3):189-98. doi: 10.2165/00007256-200636030-00001. PMID 16526831
- [Background] McMullen J, Uhl TL. A kinetic chain approach for shoulder rehabilitation. J Athl Train. 2000 Jul;35(3):329-37. PMID 16558646
- [Background] Radwan A, Francis J, Green A, Kahl E, Maciurzynski D, Quartulli A, Schultheiss J, Strang R, Weiss B. Is there a relation between shoulder dysfunction and core instability? Int J Sports Phys Ther. 2014 Feb;9(1):8-13. PMID 24567850